CLINICAL TRIAL: NCT02529826
Title: Fertility Preservation in Prepubertal Boys: An Experimental Approach
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0530-14-HMO
Record Dates: First submitted 2015-04-19; First posted 2015-08-20 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-04

CONDITIONS: Oncology [See Also, Affected System]
Keywords: Cancer-affected prepubertal boys

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Testicular biopsy (Experimental): Cancer affected prepubertal boys will undergo testicular biopsy for testicular fragments cryopreservation. The biopsy will be performed by an attending urologist, before any gonadotoxic therapy is initiated. Testicular biopsy specimens will be divided immediately on the operating table. Two thirds of the specimen will be cryopreserved for potential use by the patient at a later date and will have the patient's details and will stay at the sperm bank of Hadassah Medical Center. The other third of specimen will be used for research purposes in an effort to advance the science of isolating and culturing human SSC's for fertility research.
  Interventions: Procedure: Testicular Biopsy

INTERVENTIONS:
Procedure: Testicular Biopsy — An open testicular biopsy will be performed by an attending urologist under general anesthesia.

SUMMARY:
Due to remarkable advances in cancer treatments, the investigators are witnessing a growing population of long-term survivors of childhood malignancies. However, fertility in adult life may be severely impaired by gonadotoxic therapies. Since prepubertal boys cannot produce spermatozoa, banking of testicular tissue prior to gonadotoxic treatment is a crucial step towards fertility preservation for this population. Several centers around the world are now cryopreserving testicular tissue for prepubertal boys in anticipation that future technologies will allow the utilization of the banked samples for fertility restoration.

Testicular tissue cryopreservation has now emerged as the leading strategy for fertility preservation in prepubertal boys before gonadotoxic treatments. Fertility restoration can theoretically be obtained after allo-transplantation of testicular tissue fragments that preserve both the SSCs and the supporting microenvironment (spermatogonial stem-cell niche).

DETAILED DESCRIPTION:
As treatment regimens for pediatric oncologic malignancies have improved, more and more survivors are entering their reproductive years. Since gonadal damage is a relatively common and unfortunate consequence of the treatments used to cure pediatric cancer as well as certain hematological conditions and immunodeficiencies, maintenance of fertility is extremely important with regard to long-term quality of life for these survivors. Consideration must be given to whether a child's fertility is likely to be impacted by his or her treatment. Ideally, this should occur before the start of therapy, when a window of opportunity may exist to preserve the patient's future reproductive potential. Developments in the area of sperm banking and reproductive technologies have made it possible to offer viable options to preserve fertility to pubertal males undergoing cancer therapy. Pubertal males can produce a semen sample prior to starting gonadotoxic therapy and cryopreserve the sperm for future use. Because current methods of oocyte fertilization can utilize as few as one motile sperm, this method has proven to be successful even when the number of sperm, which are frozen, is small. Unfortunately, prepubertal males pose a particular challenge for fertility preservation. These boys cannot produce semen for cryopreservation by masturbation. They also do not have mature spermatozoa. Although the prepubertal testis does not produce mature spermatozoa, it does contain the diploid stem-germ cells from which haploid spermatozoa will be derived. For these at risk prepubertal boys, as well as for pubertal boys who may not be able to sperm bank, a recent and encouraging approach is the use of cryopreserved testicular tissue. While important strides have been made in animal research in this area, the use of testicular tissue cryopreservation in humans remains experimental. If prepubertal testicular tissue could be acquired and banked before starting gonadotoxic therapy, this tissue could then be thawed and the stored germ cells reimplanted into the patient's own testes, a procedure known as germ-cell transplantation. Alternatively, the stored cells could be matured in vitro until they can achieve fertilization by use of intracytoplasmic sperm injection (ICSI).

Research with animal models has demonstrated that there are several methods to use germ cells to obtain mature spermatozoa for fertilization including autotransplantation, and xenotransplantation. Autotransplantation is considered more acceptable than xenotransplantation, although both have been successful in mouse models. In rodents, autotransplantation has resulted in restored spermatogenesis and mice have reproduced in vivo. Investigators have demonstrated that microinjecting a crude suspension of germ cells into mice rendered sterile can restore spermatogenesis and fertility. Similar success has been reported in rats and larger mammals. Restoration of spermatogenesis is also possible with cryopreserved cells. It has been estimated that 70% of spermatogonial cells can survive after freezing and thawing. Malignant contamination remains one of the main concerns surrounding transplantation, though the few studies that address this issue are controversial in their findings. Progress in addressing this question has been made in mouse models, particularly with the use of fluorescence-activated cell sorting to negatively sort malignant cells from cell suspensions.

Because cryopreservation and transplantation of SSCs is currently successful in animals, application in humans seems likely in the near future. The possibility of infertility is an issue many families need to grapple with as they agree to initiate chemotherapy on their sons. Since this method requires testicular biopsies, both parental desire and the acceptability of SSC collection are important to assess. Recently, researchers interviewed 318 parents regarding their acceptance of such an idea. They asked parents to think hypothetically about the following scenario, "If there was an experimental procedure available at diagnosis, would you allow your sons to undergo a testicular biopsy in an attempt to collect SSCs?" At diagnosis, SSC collection by means of testicular biopsy was theoretically approved by 61% of these parents. They also observed that the desire to cryopreserve SSCs was not related to potential harmfulness of the oncological treatment, indicating that even a minor chance of infertility was considered as a major burden in respect to the ultimate quality of life. These data indicate that the translation of current animal experiments on SSC collection and transplantation into clinical care is desired by parents from prepubertal boys with cancer.

This is a novel, experimental protocol that requires collaborations between clinicians and basic scientists. There are several key clinical and translational points that have to be considered, including the beliefs and concerns of parents and prepubertal boys with cancer, the ability to perform a testicular biopsy adequately without negative sequelae, as well as tissue storage for fertility and research purposes, notably the viability of biopsy samples for downstream in vitro and functional genomics studies.

The goal of the present proposal is to develop clinical, translational, and basic science initiatives which will allow for an extensive, dedicated program for the acquisition and storage of testicular tissue from prepubertal males seen at Hadassah Medical center as well as at collaborating institutions in Israel and across the world. Developing the means for tissue distribution and handling as well as long-term tissue storage are critical components, especially since testicular tissue might be decades in storage prior to use in a fertility setting. Most importantly, a cryopreservation protocol for human testicular tissue has to be developed de novo for this initiative to ultimately become a standard option for fertility preservation for prepubertal males with cancer as well as for those with blood diseases or immunodeficiency who will be undergoing stem cell transplant.

An open testicular biopsy will be performed by an attending urologist (effort will be made to perform the procedure concurrently during a procedure when the patient is under general anesthesia for another purpose, i.e. central line placement, bone marrow aspirates/biopsies). This procedure will occur before any gonadotoxic therapy is initiated. Nevertheless, in cases of emergent chemotherapy treatment, the procedure may be done after chemotherapy since the toxicity for testicular stem cells is not known. A 10 mm incision is made in the superior pole of the testis and an approximately 5% portion of the extruded seminiferous tubules is excised (about 2 mm x 4 mm x 10 mm; approximately 1 gram of tissue). This is the size of a normal testis biopsy done for clinical reasons such as evaluation for cancer. In infants or very young boys the size of the incision and the biopsy is under the discretion of the urologist.

Testicular biopsy specimens will be divided immediately on the operating table. Two thirds of the specimen (termed Specimen #1) will be cryopreserved in Sperm Wash Media for potential use by the patient at a later date. A freezing protocol (slow freezing) currently in place for adult human testicular tissue cryopreservation will be implemented for the current proposal, and has been published in the literature for use with prepubertal testicular tissue. Specifically, 0.7 M dimethyl sulfoxide (DMSO) is used as a cryoprotective agent. Specimen #1 of the biopsy will have the patient's name, date of birth, current date, and medical record number attached. A separate sheet will also be sent with the specimen who will include phone number and current address. These specimens will stay at the sperm bank of Hadassah Medical Center.

As stated above, the other third of specimen will be used for research purposes in an effort to advance the science of isolating and culturing human SSCs for fertility research. These portions will be stripped of all personal health identifiers at the time of division and a unique identifying code will be assigned.

The risks of this study pertain to the testicular biopsy. The side effects from this procedure are mild. Pain related to the procedure is expected and is easily controlled with mild to moderate analgesic medications.

The benefit is that the patient may be able to use the frozen testicular biopsy tissue and/or cultured SSC's derived from the biopsy to preserve their fertility in the future. At this time, however, it is imperative to note that this procedure is purely experimental. The time frame for this study is defined from the date of recruitment until the date of clinical utilization of the cryopreserved tissue for fertility restoration up to forty years.

We will collect any adverse outcomes, which occur during (intra-operatively) or after the testicular biopsy including pain, bleeding and/or infection. Events will be tracked and recorded for one week after the procedure, a time frame well beyond the 2-3 day recovery time that is associated with this type of biopsy. Events clearly related to the subject's cancer or cancer treatment and not specifically to the testicular biopsy will not be collected/reported.

ELIGIBILITY:
Inclusion Criteria:

* Prepubertal males newly diagnosed with high risk malignancy (not testicular), and whose treatment will include therapy with agents that place the boy at high risk for infertility are also eligible.

Exclusion Criteria:

* None

Ages: 3 Months to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-11; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Number of cancer affected prepubertal boys who will undergo testicular cryopreservation for fertility restoration. | The time frame for this study is defined from the date of recruitment until the date of clinical utilization of the cryopreserved tissue for fertility restoration, up to forty years
  The investigators will report the number of cancer affected prepubertal boys that will undergo testicular cryopreservation for future fertility restoration.

CONTACTS AND LOCATIONS:
Overall Officials: Doron Kabiri, MD, Principal Investigator — Hadassah Hebrew Medical Center
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Derived] Kabiri D, Safrai M, Gropp M, Hidas G, Mordechai-Daniel T, Meir K, Revel A, Imbar T, Reubinoff B. Establishment of a controlled slow freezing-based approach for experimental clinical cryopreservation of human prepubertal testicular tissues. F S Rep. 2021 Nov 5;3(1):47-56. doi: 10.1016/j.xfre.2021.11.001. eCollection 2022 Mar. PMID 35386499